CLINICAL TRIAL: NCT06422923
Title: A Phase 1/2 Study of NRTX-1001 Neuronal Cell Therapy in Drug-Resistant Bilateral Temporal Lobe Epilepsy (MTLE)
Brief Title: A Phase 1/2 Study of NRTX-1001 Neuronal Cell Therapy in Drug-Resistant Bilateral Mesial Temporal Lobe Epilepsy (MTLE)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurona Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTE002
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: Bilateral Temporal Lobe Epilepsy; Bilateral MTLE; Refractory Bilateral MTLE
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): This is an open-label study of the bilateral intrahippocampal administration of NRTX-1001 in a single dose cohort of up to 10 subjects with drug-resistant bilateral MTLE.
  Interventions: Biological: NRTX-1001

INTERVENTIONS:
Biological: NRTX-1001 — Biological: NRTX-1001 is an inhibitory neural cell therapy investigational product. It is derived from a human stem cell line that has been converted into high-purity inhibitory interneurons that produce GABA. NRTX-1001 is intended to persist long-term and not require repeated administration.
  Other Names: GABA-secreting interneurons

SUMMARY:
This is a multicenter, single arm, open label clinical trial that is designed to test the safety and preliminary efficacy of single administration inhibitory nerve cells called interneurons (NRTX-1001), into both temporal lobes of subjects with drug-resistant bilateral mesial temporal lobe epilepsy.

DETAILED DESCRIPTION:
This is a multicenter, single arm, open-label study of NRTX-1001 in subjects with drug-resistant bilateral MTLE, with the objective of evaluating safety and preliminary efficacy in reducing seizure frequency. The subjects will undergo a single stereotactic CT or MRI-guided intracerebral administration of human interneurons into both temporal lobe regions of the brain. NRTX-1001 secretes the inhibitory neurotransmitter gamma-aminobutyric acid (GABA), which is intended to suppress the onset and spread of the seizures. Safety, tolerability, and effects on epilepsy disease symptoms will be assessed at approximately quarterly intervals for 2 years after the administration of NRTX-1001. After the two-year period, subjects will be followed with quarterly phone calls and annual visits in years 3 through 15.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, age 18-75 years.
2. Subjects of childbearing potential will use highly effective contraception.
3. Proven history of focal seizures of hippocampal origin with bilateral seizure foci confirmed by scalp or intracranial ictal EEG (including confirmation by recordings from responsive neurostimulation [RNS] electrodes when applicable).
4. Either

   1. bilateral hippocampal sclerosis on MRI (evidenced by increased FLAIR signal intensity in both hippocampi or by visual assessment showing reduced volume compared to normal) or
   2. bilateral temporal hypometabolism on 18-Flourodeoxyglucose Positron Emission Tomography (FDG PET) (assessed by visual assessment, comparing temporal regions to frontal/parietal lobe neocortex). In this case, ictal EEG recordings must also include intracranial confirmation.

      or
   3. a combination of unilateral instances of the evidence described in a. and b. (e.g., one side can be evidenced by criterion a. and the other side by criterion b.) MRI or PET scans used for assessment must have been acquired within 3 years of screening.
5. Subject has had at least four clinical focal seizures, including at least two clinical focal seizures with objective manifestations, on average, per month for the 6 months prior to screening.
6. Subject has previously had adequate (in opinion of investigator) therapeutic trials of at least two Anti-Seizure Medicines (ASMs).
7. Current ASM regimen, and doses of other drugs known to affect seizure frequency (e.g., antidepressants), have been stable for at least three months prior to enrollment.
8. Subject can converse and read in English or Spanish. Able to participate in required study procedures and provide signed informed consent.

Key Exclusion Criteria:

1. Epilepsy due to other and/or progressive neurologic disease.
2. Evidence of seizure focus outside hippocampus (either by seizure semiology or EEG findings).
3. MRI indicating potential malignant lesion (low-grade glioma of any type is excluded) in any location or non-malignant potentially epileptogenic lesion outside the hippocampus. Small (<2 cm) non invasive meningioma, remote from the affected temporal lobe, is not exclusionary.
4. Seizures of non-focal origin.
5. History of status epilepticus in the year prior to screening, as guided by ILAE criteria (Trinka 2015) in the judgement of the PI. A history of cluster seizures is permitted.
6. Psychogenic Non-Epileptic Seizures (PNES) within the past 3 years.
7. Severe psychiatric disorders.
8. Primary or secondary immunodeficiency.
9. Pregnancy, or currently breastfeeding.
10. Suicide attempts in past year.
11. Significant other medical conditions which would impair safe participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2042-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events at end of month 12 | 12 months after treatment

SECONDARY OUTCOMES:
Change in frequency of clinical seizures | 12 months after treatment
  Seizure frequency change during months 7-12, compared to frequency of clinical seizures in the 6-month baseline period.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Dunayevich, MD, Study Director — Neurona Therapeutics
Locations (17):
- United States (17):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Southern California Keck Hospital, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Stanford University, Palo Alto, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - SUNY Upstate Medical University, Syracuse, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - UTHealth Houston, Houston, Texas
  - UVA Health University Medical Center, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.neuronatherapeutics.com